CLINICAL TRIAL: NCT01608997
Title: Postoperative Multiparameter Outcomes During the Six Months After Rotator Cuff Repair
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0071-11-HYMC
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Shoulder Pain; Quality of Life; Satisfaction
MeSH Terms: conditions — Shoulder Pain; Personal Satisfaction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Rotator cuff tears are common amongst 50-60 year olds with no connection to their physical activity. When symptomatic, the injury affects all aspects of general health, quality of life and function. Surgical intervention is recommended only if conservative treatment fails. The purpose of the surgical intervention is to reduce pain, and improve function while improving range of motion and muscle strength around the shoulder. The purpose of the current study is to measure physical, functional, expectation, satisfaction and quality of life outcomes after rotator cuff repair surgery. Another purpose is to learn the reproducibility components of the above outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic tears in supraspinatus and infraspinatus tendon
* Symptoms of up to 12 months
* No relief from conservative treatment
* Complete or almost complete tears of up to 3cm
* Hebrew speakers

Exclusion Criteria:

* Previous trauma
* Shoulder Infection
* Recurrent dislocation
* Avascular necrosis
* Frozen shoulder
* Additional tears
* Otherwise healthy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates for rotator cuff repair due to shoulder pain and tears
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Shoulder Function | Six Months
  Outcome measurements will be collected through the use of the Quick Disability of Arm Shoulder and Hand Score (QuickDASH) questionnaire.
Quality of Life | Six Months
  Outcome measurements will be collected through the use of the Twelve Item Health Status Survey (SF12)

SECONDARY OUTCOMES:
Self-Rated Improvement, Expectations and Satisfaction | Six Months
  Outcome measurements will be collected through the use of the Patient Global Rating of Change Questionnaire
Range of Motion of the Shoulder | Six Months
  Outcome will be measured through the use of a digital inclinometer
Isometric strength around the shoulder | Six months
  Outcome will be measured by a hand-held dynamometer (HHD)

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel